CLINICAL TRIAL: NCT00948064
Title: A Phase 2 Trial of Vorinostat in Combination With Azacitidine in Patients With Newly-Diagnosed Acute Myelogenous Leukemia (AML) or Myelodysplastic Syndrome (MDS) Who Are Ineligible for Other Leukemia Protocols
Brief Title: Vorinostat in Combination With Azacitidine in Patients With Newly-Diagnosed Acute Myelogenous Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0685; NCI-2009-01495 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Leukemia
Keywords: Leukemia; Acute Myelogenous Leukemia; AML; Myelodysplastic Syndrome; MDS; Vorinostat; SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza; Azacitidine; 5-Azacitidine; 5-Aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Vorinostat; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vorinostat with Azacitidine (Experimental): ARM A: Azacitidine 75 mg/m^2/day by vein over 15 - 30 minutes daily for 5 days (Days 1 - 5). Vorinostat 200 mg by mouth three time a day with food for 5 days (Days 1 - 5). Courses repeated every 3 to 8 weeks.
  Interventions: Drug: Vorinostat; Drug: Azacitidine
- Azacitidine (Experimental): ARM B: Azacitidine 75 mg/m^2 /day by vein over 15 - 30 minutes daily for 5 days (Days 1 - 5). Courses repeated every 3 to 8 weeks.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Vorinostat — 200 mg by mouth three (3) times per day with food for 5 days (Days 1 - 5)
  Other Names: SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza
  Arms: Vorinostat with Azacitidine
Drug: Azacitidine — 75 mg/m^2/day given intravenously over 15 - 30 minutes daily for 5 days (Days 1 - 5)
  Other Names: 5-Azacitidine; 5-Aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816

SUMMARY:
The goal of this clinical research study is to learn if the combination of azacitidine and vorinostat can help to control AML or MDS better than azacitidine alone. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Azacitidine is designed to block certain genes in cancer cells whose job is to stop the function of the tumor-fighting genes. By blocking the "bad" genes, the tumor-fighting genes may be able to work better.

Vorinostat is designed to cause chemical changes in different groups of proteins that are attached to DNA (the genetic material of cells), which may slow the growth of cancer cells or cause the cancer cells to die.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups.

* If you are in Group 1, you will receive azacitidine and vorinostat.
* If you are in Group 2, you will receive azacitidine alone.

For the first 40 patients, you will have an equal chance of being in either group. After the first 40 patients, you will have a higher chance of being assigned to a group based on the results from previous participants.

Study Drug Administration:

On Days 1-5 of every cycle, you will receive azacitidine by vein over 15-30 minutes.

If you are in Group 1, you will also take vorinostat by mouth 3 times a day with food on Days 1-5 of every cycle.

If you cannot take vorinostat by mouth during a cycle, you will receive only azacitidine during that cycle. You will begin taking vorinostat by mouth again when you are able.

Your dose of study drugs may be lowered if you experience side effects.

You may receive a drug such as ondansetron before each dose of azacitidine to prevent nausea and vomiting.

If you have diarrhea, you will take a drug such as Imodium (loperamide) to prevent diarrhea.

Study Visits:

Once a week of Cycle 1, the following tests and procedures will be performed:

* Your complete medical history will be recorded.
* You will have a physical exam.
* You will be asked if you have experienced any intolerable side effects.
* Blood (about 1-2 tablespoons) will be drawn for routine tests.

On Day 28 of Cycle 1 (+/- 3 days), you will have bone marrow aspiration to check the status of the disease. To collect a bone marrow aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.

If the doctor thinks it is needed, you will have extra bone marrow aspirations during the later cycles to check the status of the disease.

One (1) time each cycle of Cycles 2 and beyond, the following tests and procedures will be performed:

* Your complete medical history will be recorded.
* You will have a physical exam.
* You will be asked if you have experienced any intolerable side effects.
* If the doctor thinks it is needed, blood (about 2 tablespoons) will be drawn for routine tests.

Length of Study:

You will be on active study for up to 12 cycles (about 12-18 months). You will be taken off study if the disease gets worse or you experience intolerable side effects.

This is an investigational study. Vorinostat is FDA approved and commercially available for the treatment of cutaneous T-cell lymphoma. Azacitidine is FDA approved commercially available for the treatment of MDS. The combination of these drugs for use in patients with intermediate-1 or higher risk MDS and AML is investigational.

Up to 80 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed AML or MDS (Intermediate 1 or higher risk)
2. Patient must have at least one of the following: a. Creatinine >/= 2 mg/dL; b. total Bilirubin >/= 2 mg/dL; c.ECOG Performance Status equal to 3 or 4; and d. is ineligible for participation on a protocol of higher priority
3. Patients must provide written informed consent.
4. Patients must be age > 18 years due to lack of safety information with these agents in children.
5. Patient agrees to: 1) Use 2 adequate methods of contraception to prevent pregnancy (either 2 barrier methods or a barrier method plus a hormonal contraceptive method) or 2) abstain from heterosexual activity throughout the study starting with Visit 1.
6. Female patients of childbearing potential should have a negative pregnancy test (serum) within 72 hrs. of study enrollment.

Exclusion Criteria:

1. Patients must not have the favorable cytogenetic abnormalities of inv (16), t (16;16), t (8;21), or t (15;17).
2. Patients receiving any anti-leukemic therapy with the exception of Hydroxyurea prior to study enrollment. Prior growth factor therapy is acceptable. Hydroxyurea could be used at the discretion of the treating physician. A single or a two day dose of cytarabine (up to 3 g/m^2) for emergency use is allowed as prior therapy.
3. Patient has a prior history of treatment with HDAC inhibitors. Patients who have received valproic acid (VPA) for the treatment of seizures may be enrolled on this study, but must not have received VPA within 30 days of study enrollment.
4. Patient is unable to take and/or tolerate oral medications on a continuous basis, examples include patients on a ventilator, or have altered mental status that precludes safe oral route of administration.
5. Patient has active hepatitis A, B, or C infection.
6. Patient is pregnant or breast-feeding.
7. Patient has a known allergy or hypersensitivity to any component of vorinostat or azacitidine.
8. History of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-09-08 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2017-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Montalban-Bravo G, Huang X, Naqvi K, Jabbour E, Borthakur G, DiNardo CD, Pemmaraju N, Cortes J, Verstovsek S, Kadia T, Daver N, Wierda W, Alvarado Y, Konopleva M, Ravandi F, Estrov Z, Jain N, Alfonso A, Brandt M, Sneed T, Chen HC, Yang H, Bueso-Ramos C, Pierce S, Estey E, Bohannan Z, Kantarjian HM, Garcia-Manero G. A clinical trial for patients with acute myeloid leukemia or myelodysplastic syndromes not eligible for standard clinical trials. Leukemia. 2017 Feb;31(2):318-324. doi: 10.1038/leu.2016.303. Epub 2016 Oct 31. PMID 27795561
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 08, 2009 to March 20, 2014. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 110 participants enrolled, 31 were enrolled in the Phase I portion of the study and 79 were enrolled in Phase II part of the study.
Groups:
- Vorinostat With Azacitidine, Phase I: Open-Label: Azacitidine 75 mg/m^2/day by vein over 15 - 30 minutes daily for 5 days (Days 1 - 5). Vorinostat 200 mg by mouth three times a day with food for 5 days (Days 1 - 5). Courses repeated every 3 to 6 weeks.
- Vorinostat With Azacitidine, Phase II: Randomized, ARM A: Azacitidine 75 mg/m^2/day by vein over 15 - 30 minutes daily for 5 days (Days 1 - 5). Vorinostat 200 mg by mouth three time a day with food for 5 days (Days 1 - 5). Courses repeated every 3 to 8 weeks.
- Azacitidine, Phase II: Randomized, ARM B: Azacitidine 75 mg/m^2 /day by vein over 15 - 30 minutes daily for 5 days (Days 1 - 5). Courses repeated every 3 to 8 weeks.
Period: Phase I
Arm/Group | Vorinostat With Azacitidine, Phase I | Vorinostat With Azacitidine, Phase II | Azacitidine, Phase II
Started | 31 | 0 | 0
Completed | 30 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — No treatment received | 1 | 0 | 0
Period: Phase II
Arm/Group | Vorinostat With Azacitidine, Phase I | Vorinostat With Azacitidine, Phase II | Azacitidine, Phase II
Started | 0 | 52 | 27
Completed | 0 | 51 | 26
Not Completed | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorinostat With Azacitidine, Phase I | Vorinostat With Azacitidine, Phase II | Azacitidine, Phase II | Total
Number analyzed (Participants) | 31 | 52 | 27 | 110
Age, Continuous [Median (Full Range); unit: years] | 74 [44 to 83] | 71 [30 to 89] | 71 [54 to 90] | 72 [44 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 9 | 33
  Male | 22 | 37 | 18 | 77
Region of Enrollment [Number; unit: participants]
  United States | 31 | 52 | 27 | 110

OUTCOME MEASURES:

1. Primary Outcome: Survival at Day 60
Description: Assessment of survival for outcome done on 60 days following therapy and includes participants alive for at least 60 days. Survival is calculated from start of therapy until death from any cause.
Time Frame: Phase I, Baseline to 60 days following first treatment.
Population: Of the 31 enrolled participants, 30 were evaluable and 1 participant never received treatment.
Measure: Number; unit: participants
Arm/Group | Vorinostat With Azacitidine, Phase I
Number analyzed (Participants) | 30
participants | 24

2. Primary Outcome: Response Rate
Description: Number of participants with Complete Response (CR) in AML requiring disappearance of all signs and symptoms related to disease, normalization of peripheral counts (absolute neutrophil count 10^9/L or more, platelet count 100 x 10^9/L or more), and a marrow with 5% or less marrow blasts; a hematologic improvement (HI) defined as a CR except for a platelet count increase by 50% to above 30 x 10^9/L. For MDS, the International Working Group criteria used to assess response.
Time Frame: 12-18 Months
Population: Out of 79 participants enrolled in Phase II, 2 participants were not evaluable - 1 participant was removed from study per treating physician discretion and the other was removed per participant's request.
Measure: Number; unit: participants
Arm/Group | Vorinostat With Azacitidine, Phase I | Vorinostat With Azacitidine, Phase II | Azacitidine, Phase II
Number analyzed (Participants) | 30 | 51 | 26
participants
  Complete Response | 9 | 11 | 8
  Hematologic Improvement | 0 | 1 | 1
  No Response | 21 | 39 | 17
  Not Evaluable | 0 | 1 | 1

3. Primary Outcome: Survival at Day 60
Description: as for outcome 1
Time Frame: Phase II, Baseline to 60 days following first treatment.
Population: Of the 79 participants enrolled, 78 were evaluable and 1 participant withdrew from study.
Measure: Number; unit: participants
Arm/Group | Vorinostat With Azacitidine, Phase II | Azacitidine, Phase II
Number analyzed (Participants) | 51 | 27
participants | 43 | 18

ADVERSE EVENTS:
Time Frame: Adverse event collected when occur within 30 days of discontinuation of dosing or completion of participation in study if the last scheduled visit occurs at a later time. Overall study period: January 2009 to April 2015.
Description: Of the 31 participants enrolled in the phase I portion of this study, 1 participant did not receive treatment; hence only 30 participants were evaluable for serious and other adverse events.
Arm/Group | Vorinostat With Azacitidine, Phase I | Vorinostat With Azacitidine, Phase II | Azacitidine, Phase II
Serious Adverse Events (participants affected / at risk) | 15/30 | 36/52 | 18/27
Other Adverse Events (participants affected / at risk) | 21/30 | 45/52 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat With Azacitidine, Phase I (N=30) | Vorinostat With Azacitidine, Phase II (N=52) | Azacitidine, Phase II (N=27)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3)
Clostridium Difficile Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 8 (8) | 11 (11) | 6 (6)
Dehydration (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Hemoptysis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 2 (3) | 1 (1)
Infection Pneumonia (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Infection Pseudomonas Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle Weakness (General disorders) | 2 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Neutropenic Fever (Infections and infestations) | 4 (6) | 9 (14) | 5 (7)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Seizures (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular Arrythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Acute Maxillary Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Altered Mental Status (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (General disorders) | 0 (0) | 4 (4) | 0 (0)
Blurry Vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Debridement of Anal Wound and Laproscopic Placement of Colostomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Deep Vein Thrombosis of Upper Extremity at PICC Site (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Elevated Bilirubin (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Emergency Surgery to Evacuate Subdural Hematoma (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Failure to Thrive (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Bleed (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Hip Prosthesis Revision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Neutropenic Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orthostatic Hypotension (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 4 (6) | 2 (2)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Renal Insufficiency/Edema (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Right Hip Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tumor Lysis Syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Weakness (General disorders) | 0 (0) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat With Azacitidine, Phase I (N=30) | Vorinostat With Azacitidine, Phase II (N=52) | Azacitidine, Phase II (N=27)
Alanine Transaminase (ALT) (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Bilirubin (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (10) | 17 (44) | 6 (13)
Creatinine (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (6) | 14 (20) | 0 (0)
Fatigue (General disorders) | 4 (4) | 34 (87) | 12 (20)
Neutropenic Fever (Infections and infestations) | 3 (8) | 8 (13) | 2 (2)
Hair Loss/Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 5 (7) | 0 (0) | 0 (0)
Mucositis/Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle Weakness (General disorders) | 1 (1) | 10 (16) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 20 (40) | 2 (3)
Opportunistic Infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 3 (8) | 2 (3)
Urinary Frequency/Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac General (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 12 (17) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 13 (26) | 0 (0)
Edema (Blood and lymphatic system disorders) | 0 (0) | 12 (19) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage/Bleeding (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 9 (12) | 0 (0)
Mental Status (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Neurology (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 3 (5) | 0 (0)
Occular/Visual (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 3 (6) | 0 (0)
Voice Changes/Dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Watery Eye (Eye disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes